CLINICAL TRIAL: NCT05567757
Title: Initial Safety Study of the TRUE AVC in Hemodialysis Access (TRUE AVC I Study)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vascudyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-002
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: End Stage Renal Disease
Keywords: hemodialysis; arteriovenous access
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Prospective, nonrandomized, single-arm, single-center, open-label, initial safety study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Investigational (Experimental): Study subjects implanted with a TRUE AVC as an arteriovenous conduit for hemodialysis
  Interventions: Biological: Arteriovenous conduit implant

INTERVENTIONS:
Biological: Arteriovenous conduit implant — Study subjects will be implanted with an arteriovenous shunt for hemodialysis access in the upper extremity

SUMMARY:
Prospective, nonrandomized, single-arm, single-center, open-label, initial safety study in subjects requiring hemodialysis. Subjects will be followed with physical evaluation and ultrasound vessel imaging at days 15, 29, 57 and weeks 12, 26. Extended follow up on patent conduits only at weeks 52 and 104.

DETAILED DESCRIPTION:
Twenty (20) patients with end-stage kidney disease (ESKD), who are poor candidates for an autogenous fistula creation and either on hemodialysis or expected to start hemodialysis within 12 weeks of study conduit implantation will be implanted with a TRUE AVC as an arteriovenous conduit in the upper extremity. Study subjects will be evaluated for implant safety and patency at 26 weeks. Subjects will be followed with physical evaluation and ultrasound vessel imaging at days 15, 29, 57 and weeks 12, 26. Extended follow up on patent conduits only at weeks 52 and 104.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with end stage kidney disease (ESKD) who are poor candidates for creation of a simple autogenous AV fistula (without requiring transposition) and therefore need placement of an AV access in the upper extremity to start or maintain hemodialysis therapy.
2. Either on hemodialysis or expected to start hemodialysis within 12 weeks of study conduit implantation.
3. Patients between 18 and 75 years old, inclusive.
4. Verify adequate arterial flow and venous runoff using duplex ultrasound and venogram. Ensure outflow vein is at least 5 mm in diameter with good compliance.
5. Hemoglobin ≥8g/dL and platelet count ≥100,000/mm3 prior to implant.
6. Other hematological and biochemical parameters within a range consistent with ESKD and acceptable for the administration of regional or general anesthesia prior to implant.
7. Adequate liver function, defined as serum bilirubin ≤1.5 mg/dL; GGT, AST, ALT, and alkaline phosphatase ≤2x upper limit of normal or INR ≤ 1.5 prior to implant.
8. Life expectancy of at least 1 year.
9. Negative COVID-19 test within 3 days prior and negative for symptoms within 14 days prior to implant.
10. Female subjects must be either:

    1. Of non-childbearing potential, which is defined as post-menopausal (at least 1 year without menses prior to Screening) or documented surgically sterile or post hysterectomy (at least 1 month prior to Screening)
    2. Or, of childbearing potential, in which case:

    i. Must have a negative urine blood pregnancy test at Screening, and ii. Must agree to use at least one form of the following birth control methods for the duration of the study:

1. Established use of oral, injectable or implanted hormonal methods of contraception 2. Placement of an intrauterine device or intrauterine system 3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/ gel/ film/ cream/ suppository 11. Able to communicate meaningfully with investigative staff and able to comply with entire study procedures.

12. Willing and competent to give written informed consent

Exclusion Criteria:

1. History or evidence of severe cardiac disease (NYHA Functional Class III or IV); myocardial infarction within six months prior to study entry; ventricular tachyarrhythmias requiring continuing treatment; unstable angina; or ejection fraction < 50%.
2. Uncontrolled or poorly controlled diabetes defined as A1C > 8; hospitalization for poor glucose control within the previous 6 months.
3. History or evidence of severe peripheral vascular disease in the upper limbs
4. Known or suspected central vein obstruction on the side of planned study conduit implantation. Avoid patients with current subclavian catheters or leads on the side of the study conduit implant. If the patient had previous subclavian catheters or leads on the implant side, verify adequate runoff with a venogram.
5. Documented hypercoagulable state or history of thromboembolic events or history of repeated venous catheter clotting.
6. Known Positive COVID 19 test result or known exposure to COVID 19 in past 3 months.
7. Known active infection including dental infection, osteomyelitis and other conditions which could present a local or systemic risk of infection.
8. Bleeding diathesis.
9. Contraindication to or known serious allergy to anticoagulant, aspirin, or planned antiplatelet therapy. History of heparin-induced thrombocytopenia.
10. Immunodeficiency including AIDS / HIV or active autoimmune disease, or on immunosuppressant therapy.
11. Autoimmune nephropathy
12. Previous PTFE graft in the operative limb unless the TRUE AVC can be placed more proximally than the previous failed graft.
13. More than 1 failed PTFE graft in the operative limb.
14. Patients receiving an AV access which crosses the elbow.
15. Patients receiving a lower extremity AV access.
16. Treatment with any investigational drug or device within 60 days prior to study entry or ongoing participation in a clinical trial of an investigational product.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-report of gender identity
Enrollment: 11 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Adverse Event Incidence | through 26 weeks post implant
  incidence of clinically significant aneurysm, anastomotic bleeding, study conduit or anastomotic rupture, study conduit infection, and implant site irritation, inflammation, or infection
Patency | through 26 weeks post implant
  Kaplan-Meier freedom from loss of primary patency, primary assisted patency, and secondary patency.

SECONDARY OUTCOMES:
Change in antigen sensitivity | baseline through 4 weeks
  Assess changes in anti-HLA sensitivity in each implant recipient, from baseline through four weeks, using panel reactive antibody (PRA) test
Rate of Interventions | 26 weeks
  Rate of interventions needed to maintain patency

CONTACTS AND LOCATIONS:
Overall Officials: Ernesto Alvarado, MD, Principal Investigator — Centro de Asistencia Renal, Río Hato, Coclé, Panamá
Locations (1):
- Centro de Asistencia Renal, Río Hato, Provincia de Coclé, Panama